CLINICAL TRIAL: NCT02256579
Title: Vietnam-Japan Cooperative Research on Prognosis of HIV-1-infection -Clinical Utility of Urinary beta2 Microglobulin as an Early Marker of Renal Dysfunction Caused by Use of Tenofovir in Vietnamese HIV-Infected Patients-
Brief Title: Utility of Urinary beta2 Microglobulin as an Early Marker of Renal Dysfunction in Vietnamese HIV-Infected Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Center for Global Health and Medicine, Japan (Other Government)
Responsible Party: Sponsor
Other Study IDs: NCGM-G-001074-01
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infection; Renal Function Disorder; Renal Tubular Disorder
Keywords: TDF:Tenofovir, Urine beta2microglobulin
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Complete blood cell count, CD4+ cell count, AST, ALT, Serum-creatinine, HIV-1 plasma viral loads, HBs antigen, anti-HBc antibody, anti-HBs antibody, anti-HCV antibody, Urine-protein, Urine-creatinine and urine beta2microglobulin.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to investigate clinical utility of beta2 microglobulin as an early marker for renal dysfunction caused by Tenofovir in Vietnamese HIV-infected patients.

DETAILED DESCRIPTION:
An observational study to investigate clinical utility of beta2 microglobulin as an early marker for renal dysfunction caused by Tenofovir in Vietnamese HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients in the NHTD -ACC cohort who are under cART or will start cART and can provide written informed consents.

Exclusion Criteria:

* HIV-infected patients who drop out of treatment within 6 months from the entry.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vietnamese HIV-infected patients who are registered in the NHTD (National Hospital of Tropical Diseases) -ACC (AIDS Clinical Center, NCGM) cohort.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-11 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of urinary beta2microglobulin, urinary protein and serum creatinine among Vietnamese HIV-infected patients | 3 years
  Follow up Vietnamese HIV-infected patients, for their renal function including urinary beta2microglobulin, urinary protein and serum creatinine for 3 years

SECONDARY OUTCOMES:
Evaluation of risk factors for renal dysfunction and tubular dysfunction | 3 years
  Risk factors for renal and tubular dysfunction were evaluated.
  Risk factors including:
  Age, sex, body weight, history of ART, AIDS or non-AIDS complication and concomitant use of cotrimoxazole, Hepatitis C virus antibody and Hepatitis B virus Ag antigen, CD4 positive cell count and HIV viral load.

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Oka, MD. PhD, Principal Investigator — National Center for Global Health and Medicine